CLINICAL TRIAL: NCT03923647
Title: Laparoscopic Exploration Versus Abdominal CT Scanning in Abdominal Trauma
Brief Title: Laparoscopic Exploration Versus Abdominal CT Scan
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Usama Amer, Usama Amer Mohammed, principal investigator, Assiut University
Other Study IDs: Laparoscopy in abd trauma
Record Dates: First submitted 2019-04-06; First posted 2019-04-22 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Penetrating Abdominal Trauma
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Laparoscopy and CT scan: Usage of laparoscopy after inflation of co2 infra umbilical
  Interventions: Device: Laparoscopy

INTERVENTIONS:
Device: Laparoscopy — Laparoscopic insertion with carbon dioxide via open technique at the umbilicus

SUMMARY:
Evaluate the efficacy and safety of laparoscopy and it's role with blunt abdominal trauma

DETAILED DESCRIPTION:
Evaluate the role of laparoscopy and Abdominal Ct scan in diagnosis and treatment of abdominal trauma and which is more effective and safe laparoscopy or CT

ELIGIBILITY:
Inclusion Criteria:

* stable patients with definite occurrence of intra-abdominal injury
* patients with equivocal result by clinical and radiological evaluation

Exclusion Criteria:

* patients with penetrating abdominal trauma
* stable patients not in need for any intervention for conservative management
* patients with marked haemodynamic instability
* polyt-traumatized Patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable patients with abdominal trauma with good general conditions
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Evaluate the role of laparoscopy in diagnosis and management of abdominal trauma | Baseline
  Evaluate the efficacy and safety of laparoscopy in diagnosis of abdominal trauma in comparison to abdominal CT scanning in 30 stable patients with with abdominal trauma
Evaluate the role of Abdominal CT scanning in diagnosis of abdominal trauma | Baseline
  Evaluate the accuracy of CT scanning in diagnosis of abdominal trauma according to 1- age of the patient 2- amount of dye 3- general conditions of the patient 4- history of medical disease